CLINICAL TRIAL: NCT02625675
Title: Using Thoracic Ultrasound to Predict Pleurodesis Success in Malignant Pleural Effusions: a Pilot Study
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: TUS Pleurodesis
Record Dates: First submitted 2015-10-21; First posted 2015-12-09 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Malignant Pleural Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Ultrasound scan

SUMMARY:
The observational pilot study at the Churchill Hospital, funded by Oxford Respiratory Trials Unit, will assess the feasibility and efficacy of thoracic ultrasound (TUS) assessment in patients undergoing talc pleurodesis via intercostal chest drain (ICD) for recurrent symptomatic malignant pleural effusions (MPE). Participants will undergo TUS pre and post pleurodesis on up to four occasions. We hypothesise that a TUS scoring system will be able to predict short and long-term pleurodesis success earlier than current conventional medical practice allows. This study may ultimately allow the proposal of a treatment algorithm to manage patients with MPE in a more efficient manner.

ELIGIBILITY:
Inclusion Criteria:

* The participant is willing and able to give informed consent for participation in the study.
* Adult male or female, aged 18 years or above.
* Diagnosed with a malignant pleural effusion requiring intercostal chest drain insertion and subsequent talc slurry pleurodesis for symptom relief and/or other therapeutic purposes as part of routine clinical care.

Exclusion Criteria:

* Age less than 18 years.
* Inability to provide informed consent
* Known hypersensitivity/allergy to medical talc, or other contraindication to the administration of intrapleural talc, as determined by the responsible clinician.
* Evidence of significant trapped lung that would prevent pleurodesis being performed, as determined by the clinician responsible for assessing the patient.
* Expected survival of less than one month due to underlying co-morbidities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing drainage of a malignant pleural effusion and subsequent talc pleurodesis via an intercostal chest drain as part of their routine planned care.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Clinico-radiological confirmation of pleurodesis success post pleurodesis. | 1 month
  Pleurodesis success confirmed as no radiographic and/or ultrasonographic evidence of significant pleural fluid recurrence; and/or no clinical need for further pleural intervention for symptomatic relief.
Clinico-radiological confirmation of pleurodesis success post pleurodesis. | 3 months
  Pleurodesis success confirmed as no radiographic and/or ultrasonographic evidence of significant pleural fluid recurrence; and/or no clinical need for further pleural intervention for symptomatic relief.

SECONDARY OUTCOMES:
Difference (in days) between hypothetical discharge date based on thoracic ultrasound findings and actual discharge date based on standard clinical care. | Through study completion, an average of 3 months.
Patient satisfaction with thoracic ultrasound as measured using a Likert-type scale | Through study completion, an average of 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Respiratory Trials Unit, Churchill Hospital, Oxford, United Kingdom

REFERENCES:
- [Derived] Corcoran JP, Hallifax RJ, Mercer RM, Yousuf A, Asciak R, Hassan M, Piotrowska HE, Psallidas I, Rahman NM. Thoracic Ultrasound as an Early Predictor of Pleurodesis Success in Malignant Pleural Effusion. Chest. 2018 Nov;154(5):1115-1120. doi: 10.1016/j.chest.2018.08.1031. Epub 2018 Sep 20. PMID 30243566